CLINICAL TRIAL: NCT02935010
Title: Efficacy of Antibiotic Susceptibility-based Tailored Versus Empiric Therapy for Helicobacter Pylori First-line Treatment：a Randomized Clinical Trial
Brief Title: Tailored Versus Empiric Therapy for Helicobacter Pylori Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hong Lu, MD, Doctor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: rjkls2016110
Record Dates: First submitted 2016-10-11; First posted 2016-10-17 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Bismuth quadruple therapy; Tailored therapy; Empiric therapy; clarithromycin susceptibility
MeSH Terms: interventions — Esomeprazole; Amoxicillin; Clarithromycin; Metronidazole; Levofloxacin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tailored therapy (Experimental): After antimicrobial susceptibility testing of Helicobacter pylori from biopsy samples, according to antibiotic resistance pattern of each one, give esomeprazole 20mg bid and two sensitive ones of amoxicillin,clarithromycin, metronidazole,and levofloxacin. All regimens will be given for 14 days.
  Interventions: Drug: Esomeprazole; Drug: Bismuth Potassium Citrate; Drug: Amoxicillin; Drug: Clarithromycin; Drug: Metronidazole; Drug: Levofloxacin
- Empiric therapy (Active Comparator): give esomeprazole 20mg bid, bismuth potassium citrate 600mg bid, amoxicillin 1000mg tid and metronidazole 400mg tid for 14 days
  Interventions: Drug: Esomeprazole; Drug: Bismuth Potassium Citrate; Drug: Amoxicillin; Drug: Metronidazole

INTERVENTIONS:
Drug: Esomeprazole — proton pump inhibitor
Drug: Bismuth Potassium Citrate — Gastric mucosal protective drug with anti-H. pylori effect
Drug: Amoxicillin — antibiotic for H. pylori eradication
Drug: Clarithromycin — antibiotic for H. pylori eradication
  Arms: Tailored therapy
Drug: Metronidazole — antibiotic for H. pylori eradication
Drug: Levofloxacin — antibiotic for H. pylori eradication
  Arms: Tailored therapy

SUMMARY:
With markedly increased antibiotic resistance and unsatisfactory efficacies of common empiric eradication regimens in the mainland of China, tailored therapy may be the best choice to achieve good efficacy. This study compared the eradication rates, safety, and compliance of antibiotic sensitivity-based tailored therapy compared with empiric bismuth quadruple therapy in the naive patients with Helicobacter pylori infection.

ELIGIBILITY:
Inclusion Criteria:

* Participants with non-ulcer functional dyspepsia or scarred peptic ulcer disease
* Ability and willingness to participate in the study and to sign and give informed consent
* confirmed H. pylori infection

Exclusion Criteria:

* Previous H. pylori eradication therapy
* Less than 18 years old
* With history of H. pylori infection treatment
* With previous gastric surgery
* Major systemic diseases
* Pregnancy or lactation
* Allergy to any of the study drugs
* Administration of antibiotics, bismuth, antisecretory drugs in 8 weeks prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2017-02-05 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | Six weeks after completion of therapy
  Six weeks after completion of therapy, H. pylori eradication was assessed by ¹³C-urea breath test. Eradication was defined as negative result from urea breath test (<4‰) (4‰ as the cutoff value).

SECONDARY OUTCOMES:
Rate of adverse effects | within 7 days after completion of therapy
  During the 14-day treatment period, the subjects kept a diary to score any possible side effects or discomforts. The subjects were asked to grade the severity of adverse events according to their influence on daily activities, experienced as "mild" (transient and well tolerated), "moderate" (causing discomfort and partially interfering with daily activities), or "severe" (causing considerable interference with daily activities). The side effect score recorded was based on the most severe event.
Compliance rate | within 7 days after completion of therapy
  Compliance was deﬁned as poor when they had taken less than 80% of the total medication.

OTHER OUTCOMES:
Medical cost per patient of tailored or empiric therapy | two months after completion of therapy
Ratio of medical cost to H. pylori eradication rate of each therapy | two months after completion of therapy
Ratio of incremental medical cost to incremental H. pylori eradication rate of tailored compared with empiric therapy | two months after completion of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Hong Lu, M.D., Study Chair — Renji Hospital, School of Medicine, Shanghai Jiao Tong University; Yunwei Sun, M.D., Principal Investigator — Ruijin Hospital; Hong Gao, M.D., Principal Investigator — Fudan University; Yan Zhao, M.D., Principal Investigator — Shanghai Tenth People's Hospital, Tongji University; Gang Xu, M.D., Principal Investigator — Shanghai General Hospital, Shanghai First People's Hospital, Shanghai Jiao Tong University
Locations (5):
- China (5):
  - Ruijin Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai First People's Hospital, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Tongji University, Shanghai, Shanghai Municipality
  - Zhongshan Hospital,Fudan University, Shanghai, Shanghai Municipality
  - Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-08): https://cdn.clinicaltrials.gov/large-docs/10/NCT02935010/Prot_SAP_000.pdf